CLINICAL TRIAL: NCT04247282
Title: A Sequential Window of Opportunity Trial of Anti-PD-L1/TGF-beta Trap (M7824 ) Alone and in Combination With TriAd Vaccine, and N-803 for Resectable Head and Neck Squamous Cell Carcinoma Not Associated With Human Papillomavirus Infection.
Brief Title: Anti-PD-L1/TGF-beta Trap (M7824) Alone and in Combination With TriAd Vaccine and N-803 for Resectable Head and Neck Squamous Cell Carcinoma Not Associated With Human Papillomavirus Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoyoung M. Maeng, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200024; 20-C-0024
Record Dates: First submitted 2020-01-25; First posted 2020-01-30 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms
Keywords: Immuno-oncology; Neoadjuvant Treatments; Non-HPV; Immunotherapy; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — bintrafusp alfa protein, human; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) (Experimental): M7824 (Days 1, 15)
  Interventions: Drug: M7824
- Arm B, Cohort 1 M7824 + TriAd Vaccine (ETBX-011, ETBX-051 & ETBX-061) (Day 1) (Experimental): M7824 + TriAd vaccine (ETBX-011, ETBX-051 and ETBX-061) (Days 1)
  Interventions: Drug: M7824; Biological: TriAd vaccine
- Arm C, Cohort 1 M7824 + TriAd Vaccine (Day 1) + N-803 (Day 1) (Experimental): M7824 + TriAd vaccine (Day 1) + N-803 (Day 1)
  Interventions: Drug: M7824; Drug: N803; Biological: TriAd vaccine

INTERVENTIONS:
Drug: M7824 — M7824 (1200 mg) will be administered intravenously on day 1 and 15 to patients enrolled in arm 1-3 (all three arms).
  Other Names: bintrafusp alfa
Drug: N803 — N-803 (15 mcg/kg, subcutaneously) will be given on day 1 to patients enrolled in arm 3.
  Other Names: Anktiva
  Arms: Arm C, Cohort 1 M7824 + TriAd Vaccine (Day 1) + N-803 (Day 1)
Biological: TriAd vaccine — TriAd vaccine (5 x 10e(11) viral particles (VP); subcutaneous injection) will be given on day 1 to patients enrolled in arm 2 and arm 3
  Other Names: ETBX-011, ETBX-051 & ETBX-061
  Arms: Arm B, Cohort 1 M7824 + TriAd Vaccine (ETBX-011, ETBX-051 & ETBX-061) (Day 1); Arm C, Cohort 1 M7824 + TriAd Vaccine (Day 1) + N-803 (Day 1)

SUMMARY:
Background:

Some people who get head and neck cancer will need surgery to treat their cancer. Research suggests that immunotherapy drugs may help fight head and neck cancer if given before surgery. In most cases, there is enough time between cancer diagnosis and surgery to test immunotherapy drugs. In this study, researchers are testing the safety and anti-cancer abilities of 3 drugs given before surgery for head and neck cancer.

Objective:

To learn if giving M7824 alone, or with the TriAd Vaccine (ETBX-011, ETBX-051 & ETBX-061), or with TriAd vaccine plus Anktiva (N-803) can shrink previously untreated head and neck tumors before surgery or stop the tumors from coming back after all treatment.

Eligibility:

People age 18 and older who have a head and neck cancer that has not been treated before, and the tumor must be removed with surgery.

Design:

Participants will be screened in a separate protocol.

Participants will have the following tests:

* medical history and physical exams
* computed tomography or magnetic resonance imaging scans
* tumor, mucosa, and skin biopsies
* electrocardiograms to monitor heart activity
* endoscopies (a tube is inserted through the nose to see the upper airway)
* blood and urine tests.

All participants will get bintrafusp alfa (M7824) through an intravenous infusion. For this, a small plastic tube is put into an arm vein. Some may also get the TriAd vaccine. It is injected under the skin on the arms or legs. Some may also get N-803. It is injected under the skin on the stomach.

Participants will have clinic visits while they are getting treatment and after treatment ends.

After treatment ends, participants will have their scheduled surgery. There will be two follow up visits at the National Institutes of Health (NIH) after your surgery. They will be contacted by phone or email every 2 weeks for 3 months. Then they will be contacted every 3 months for 2 years.

...

DETAILED DESCRIPTION:
Background:

* Approximately 50% of patients with advanced, non-human papilloma virus (HPV) associated head and neck squamous cell carcinoma (HNSCC) will develop locoregional or distant relapse within two years of completing definitive standard-of-care treatment.
* Two ongoing clinical trials investigating neoadjuvant programmed cell death protein 1 (PD-1) blockade before surgical resection of HNSCC suggest that immunotherapy can both cytoreduce existing disease before surgery and reduce the risk of locoregional or distant disease relapse after surgery.
* Preliminary data from these studies suggest neoadjuvant treatments can be administered without delaying planned surgical intervention.
* Experiments conducted by the Laboratory of Tumor Immunology and Biology (LTIB) demonstrated synergistic activity with tumor-targeted adenoviral vaccine plus bintrafusp alfa (M7824) plus Anktiva (N-803) in humanized mice bearing human carcinomas and in vitro studies.
* M7824 is a bifunctional fusion protein consisting of an anti-programmed death ligand 1(PD-L1) antibody and the extracellular domain of transforming growth factor beta (TGF-beta) receptor type 2, a TGF-beta trap.
* Adenoviral vaccines targeting known shared tumor antigens can generate antigen-specific T cells.
* N-803 is an interleukin 15 (IL-15)/interleukin 15 receptor (IL-15R) alpha super agonist complex that can enhance both natural killer (NK) cell and T cell anti-tumor activity via expansion and activation.
* Activity observed with neoadjuvant anti-PD-1 agents alone provides rationale for testing of M7824 alone and in combination with other immune-oncologic agents that have been shown to work in concert with M7824 in preclinical studies.
* Analysis of pre- and post-treatment tissues from HNSCC patients presents a unique opportunity to interrogate the effects the above treatment(s) on tumor.
* A dose escalation of N-803 in combination with a flat dose of M7824 was conducted at the National Cancer Institute. Thirteen patients have been treated with the combination. No dose limiting toxicities (DLTs) were observed.

Objectives:

-Determine the rate of pathologic complete response (pCR) or clinical-to-pathological downstaging in patients with previously untreated intermediate/high risk, non-HPV associated, squamous cell carcinoma of the head and neck (T1-T4, N0-N3, M0 stage II, III or IV) who receive any of the three proposed treatments: M7824 alone, M7824 plus TriAd vaccine, or M7824 plus TriAd vaccine plus N803 prior to definite surgery.

Eligibility:

* Patients must have histologically or cytologically confirmed, previously untreated intermediate/high risk, p16-negative (if oropharyngeal), squamous cell carcinoma of the head and neck (T1-T4, N0-N3, M0 stage II, III or IV)
* Men or Women; Age greater than or equal to 18 years
* Eastern Cooperative Oncology Office (ECOG) performance status less than or equal to 1

Design:

* This protocol is a sequential window of opportunity trial of Anti-PD-L1/TGF-beta trap (M7824) alone and in combination with TriAd Vaccine (ETBX-011, ETBX-051 & ETBX-061) and N-803 for non-HPV associated resectable Head and Neck Squamous Cell Carcinoma (HNSCC).
* Patients will be referred to the National Institutes of Health (NIH) for this immunotherapy treatment from surrounding academic medical centers and private physicians.
* Upon referral to the NIH, patients will be rapidly screened, and enrolled on the protocol, if appropriate.
* This trial will enroll patients in three arms sequentially to permit safety evaluation before adding the next agent.
* In the first arm of 12 patients, M7824 (1200 mg) will be administered intravenously on day 1 and 15.
* If no safety concerns, accrual will proceed to the 2nd arm, and 12 patients will enroll with M7824 (1200mg; intravenous) treatment on day 1 and 15 and TriAd vaccine (5 x 10 (11) viral particles (VP; subcutaneous) treatment on day 1 only.
* If no safety concerns, accrual will proceed to the 3rd arm, and 12 patients will enroll with M7824 ((1200mg; intravenous) treatment on day 1 and 15 plus TriAd vaccine (5 x 10(11) VP; subcutaneous injection) and N-803 (15mcg/kg, subcutaneously) treatment on day 1.
* After obtaining pre-treatment biopsies, imaging and blood collection, patients will receive the neoadjuvant immunotherapy at the NIH Clinical Center.
* Patients will then be sent back to their referring providers for their definitive standard of care surgery and adjuvant therapy as indicated based upon pathologic analysis of the surgical specimen. National Cancer Institute (NCI) investigators will have no role in directing the ensuing standard of care surgeries performed at outside institutions.
* For consistency in pathologic analysis of resection specimens, tissue blocks and/or slides will be obtained from outside institutions and be reviewed by the NCI Laboratory of Pathology.
* It is expected that up to 20 patients may enroll in one year. Thus, with 3 arms of 12 patients apiece, up to 36 evaluable patients may enroll. Accrual is expected to be completed within 2 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed, previously untreated intermediate/high risk, p16-negative (if oropharyngeal primary tumor), squamous cell carcinoma of the head and neck (T1-T4, N0-N3, M0 stage II, III or IV).
* Male or female; Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG performance status less than or equal to 1.
* Prothrombin time (PT) and partial thromboplastin time (PTT) within normal institutional limits. Patients with prolonged PTT determined to be due to lupus anticoagulant will not be excluded.
* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1000/mcL
  * Platelets greater than or equal to 100,000/mcL
  * Hemoglobin greater than or equal to 10.0 g/dL
  * Total bilirubin within normal institutional limits; in patients with Gilbert's, less than or equal to 3.0 mg/dL
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to 3X upper limit of normal.
  * Creatinine within 1.5X upper limit of normal institutional limits
* The effects of M7824, TriAd Vaccines (ETBX-011, ETBX-051 & ETBX-061), and Anktiva (N-803) on the developing human fetus are unknown. For this reason, men and women of child-bearing capacity must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study and maintain such contraception until 2 months following the last dose of any study agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document
* Patients with successfully treated hepatitis C virus (HCV) are eligible if HCV viral load is undetectable.

EXCLUSION CRITERIA:

* Patients who are immunocompromised as follows:

  * Human immunodeficiency virus (HIV) positive patients not on or not compliant with appropriate anti-retroviral therapy, patients with newly diagnosed (i.e., < 6 months) HIV, patients with an HIV viral load exceeding 400 copies/mL, HIV+ patients with a cluster of differentiation 4 (CD4) count < 150 cells/L, and HIV+ patients on antiretroviral therapy < 1 month are excluded. HIV-positive patients will also be excluded if the principal investigator (PI) determines that there is a clinically significant drug-drug interaction.
  * Chronic administration (defined as daily or every other day for continued use >14 days) of systemic corticosteroids or other immune suppressive drugs, within 14 days before treatment on study. Physiologic daily dosing of steroids is allowed. Nasal, or inhaled steroid, topical steroid creams and eye drops for small body areas are allowed.
  * Patients who have undergone allogeneic peripheral stem cell transplantation, or solid organ transplantation requiring immunosuppression
* Pregnant women are excluded from this study because M7824 is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M7824 breastfeeding should be discontinued if the mother is treated with M7824. These potential risks may also apply to other agents used in this study.
* Patients with active systemic autoimmune disease, except patients with type 1 diabetes mellitus, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring current immunosuppression, or with other endocrine disorders on replacement hormones, are not excluded if the condition is well controlled.
* Patients with a history of inflammatory bowel disease
* Patients with a history inflammatory lung disease/interstitial lung disease/pulmonary fibrosis will be excluded. Patients with clinical findings (e.g., imaging) that are suggestive of inflammatory lung disease even if not experiencing symptoms of the disorder.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents to be used in the cohort the subject will be enrolled into.
* Known allergy to eggs, egg products, aminoglycoside antibiotics (for example, gentamicin or tobramycin). Patients enrolling on the M7824 only arm will be exempt from this exclusion.
* Patients with a history of bleeding diathesis or recent clinically significant bleeding events considered by the Investigator as high risk for investigational drug treatment are excluded.
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial (including the long-term follow-up), or would interfere with the evaluation of the trial endpoints.
* Patients with prior live vaccine, investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to enrollment. Locally approved coronavirus disease (COVID) vaccines are permitted.
* Uncontrolled intercurrent acute or chronic illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (>New York Heart Association Class I), hepatic disease, unstable angina pectoris, serious cardiac arrhythmia, requiring medication, uncontrolled hypertension (systolic blood pressure (SBP>170/ diastolic blood pressure (DBP>105) or psychiatric illness/social situations within 12 months that would limit compliance with study requirements.
* Patients who have undergone major surgery within 4 weeks prior to enrollment. A biopsy will not preclude a patient from starting study.
* Patients with a history of hepatitis B (HBV) are excluded due to potential risk for viral reactivation and resulting liver injury in persons with latent HBV.
* Patients with treated or active brain metastases are not eligible because we are enrolling non-metastatic head and neck cancer patients in this trial. Standard of care treatment is different for head and neck cancer patients with and without metastatic disease.
* Subjects unwilling to accept blood products as medically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All large- scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Result] Redman JM, Donahue RN, Steinberg SJ, Marte JL, Cordes L, Floudas CS, Prins D, Turkbey EB, Soon-Shiong P, Schlom J, Gulley JL, Allen CT. Tri-Ad5 vaccine plus bintrafusp alfa for newly diagnosed, advanced-stage head and neck cancer not associated with human papillomavirus infection. Oncologist. 2025 Mar 10;30(3):oyaf006. doi: 10.1093/oncolo/oyaf006. PMID 40156838
- [Derived] Redman JM, Friedman J, Robbins Y, Sievers C, Yang X, Lassoued W, Sinkoe A, Papanicolau-Sengos A, Lee CC, Marte JL, Turkbey E, Mydlarz W, Joshi A, London NR Jr, Pierce M, Taylor R, Hong S, Nguyen A, Soon-Shiong P, Schlom J, Gulley JL, Allen CT. Enhanced neoepitope-specific immunity following neoadjuvant PD-L1 and TGF-beta blockade in HPV-unrelated head and neck cancer. J Clin Invest. 2022 Sep 15;132(18):e161400. doi: 10.1172/JCI161400. PMID 35727629
- [Derived] Saint A, Van Obberghen-Schilling E. The role of the tumor matrix environment in progression of head and neck cancer. Curr Opin Oncol. 2021 May 1;33(3):168-174. doi: 10.1097/CCO.0000000000000730. PMID 33720067
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0024.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A, Cohort 1 Bintrafusp Alfa (M7824) 1200 mg (Days 1, 15): Phase I/II M7824 (Days 1, 15)
  M7824: M7824 (1200 mg) will be administered intravenously on day 1 and 15 to patients enrolled in arm 1-3 (all three arms).
- Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1): Phase I/II M7824 + TriAd vaccine (ETBX-011, ETBX-051 and ETBX-061) (Days 1)
  M7824: M7824 (1200 mg) will be administered intravenously on day 1 and 15 to patients enrolled in arm 1-3 (all three arms).
  TriAd vaccine: TriAd vaccine (5 x 10e(11) viral particles (VP); subcutaneous injection) will be given on day 1 to patients enrolled in arm 2 and arm 3
- Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1): Phase I/II No participants were enrolled on Arm C, Cohort 1.
  M7824 + TriAd vaccine (Day 1) + N-803 (Day 1)
  M7824: M7824 (1200 mg) will be administered intravenously on day 1 and 15 to patients enrolled in arm 1-3 (all three arms).
  N803: N-803 (15 mcg/kg, subcutaneously) will be given on day 1 to patients enrolled in arm 3.
  TriAd vaccine: TriAd vaccine (5 x 10e(11) viral particles (VP); subcutaneous injection) will be given on day 1 to patients enrolled in arm 2 and arm 3
- Enrolled But Not Treated: Participant was enrolled but not treated.
Period: Overall Study
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) 1200 mg (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1) | Enrolled But Not Treated
Started | 14 | 6 | 0 | 1
Completed | 14 | 5 | 0 | 0
Not Completed | 0 | 1 | 0 | 1
Not completed — Participant declined to participate before treatment started. | 0 | 0 | 0 | 1
Not completed — Refused further treatment | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristic data collected for one participant that was enrolled but not treated is reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) 1200 mg (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1) | Enrolled But Not Treated | Total
Number analyzed (Participants) | 14 | 6 | 0 | 1 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0 | 0
  Between 18 and 65 years | 8 | 3 |  | 1 | 12
  >=65 years | 6 | 3 |  | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.54 (13.38) | 60.3 (18.41) |  | 48 (0) | 59.2 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 |  | 0 | 11
  Male | 8 | 1 |  | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 |  | 0 | 3
  Not Hispanic or Latino | 13 | 4 |  | 1 | 18
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0
  Asian | 0 | 1 |  | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0
  Black or African American | 1 | 1 |  | 0 | 2
  White | 13 | 4 |  | 1 | 18
  More than one race | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 |  | 1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience a Pathologic Complete Response (pCR)
Description: Resected tumors were reviewed one month after being on study to determine a pCR, defined as absence of malignant cells in the resected tumor specimen. A pathologist examines tumor specimens to look for malignant cells.
Time Frame: Post treatment after on study, approximately one month
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15): Phase I/II M7824 (Days 1, 15)
  M7824: M7824 (1200 mg) will be administered intravenously on day 1 and 15 to patients enrolled in arm 1-3 (all three arms).
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
Participants | 0 | 0 |

2. Primary Outcome: Number of Participants Who Experience Clinical to Pathologic Downstaging Upon Analysis of Resected Tumor After Completing Study Treatments
Description: Clinical-to-pathologic downstaging is when the numerical pathological stage is lower than the initial numerical clinical stage (i.e., II to I)
Time Frame: up to 4 months after enrollment
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
Participants | 6 | 2 |

3. Secondary Outcome: Proportion of Participants With a Complete Response (CR) + Partial Response (PR) Measured by Computed Tomography (CT) Imaging and the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Response was measured by CT imaging and the RECIST to determine whose tumors shrunk after therapy. CR is disappearance of all target lesions, and PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 21-28 days from enrollment, up to a maximum of 28 days
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started.
Measure: Number; unit: proportion of participants
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
proportion of participants | 0 | 0 |

4. Secondary Outcome: Number of Participants That Experienced Grade 3 or 4 Immune Related Adverse Events (irAEs)
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 3 is severe. Grade 4 is life-threatening. Permanent treatment discontinuation is required in some cases of immune-related Grade 4 AEs (e.g., Grade 4 rash/inflammatory dermatitis, nephritis,..). Permanent treatment discontinuation is not required when the AE is manifested by a single laboratory value out of normal range without any clinical correlates.
Time Frame: 2 weeks
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
Participants
  Grade 3 Vasculitis | 1 | 0 |
  Grade 4 Pneumonitis | 0 | 1 |

5. Secondary Outcome: Probability of Being Alive and Recurrence Free
Description: Probability of being alive and recurrence (disease) free after treatment reported along with 95% confidence intervals. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, Disease recurrence is defined as the cancer comes back evidenced by imaging, clinical exam and/or biopsy.
Time Frame: 1 and 2 years
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
percent probability
  1 year | 84.6 [51.2 to 95.9] | 83.3 [27.3 to 97.5] |
  2 years | 84.6 [51.2 to 95.9] | 83.3 [27.3 to 97.5] |

6. Secondary Outcome: Percentage of Participants Who Are Alive
Description: Participants who are alive after therapy reported along with a 95% confidence interval.
Time Frame: Participants were followed to see if they were alive and recurrence free for up to 2 years from study enrollment.
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started. The data reported is observed data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
percentage of participants
  1 year | 92.3 [56.6 to 98.9] | 83.3 [27.3 to 97.5] |
  2 years | 84.6 [51.2 to 95.9] | 83.3 [27.3 to 97.5] |

7. Secondary Outcome: Number of Participants With Treatment-related Adverse Events Causing a Delay of 4 Weeks or More Beyond Planned Surgery
Description: Here is the number of participants with treatment-related adverse events causing a delay of 4 weeks or more beyond planned surgery. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: 4 weeks or more beyond surgery, up to 2 years
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
Participants | 0 | 0 |

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 2 years and 12 days for Arm A, and 2 months and 29 days for Arm B.
Population: 20/21 participants were analyzed because one participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
Number analyzed (Participants) | 14 | 6 | 0
Participants | 14 | 6 |

ADVERSE EVENTS:
Time Frame: All adverse events (AEs), including clinically significant abnormal findings on laboratory evaluations, regardless of severity, will be followed until return to baseline or stabilization of event. From first study intervention day 1 to 30 days after participant received the last product administration. After 90 days, only adverse events grade ≥3 & possibly related to the study investigational agent need to be recorded. Approximately 2 years & 12 days for Arm A, and 2 months & 29 days for Arm B.
Description: 20/21 participants were analyzed because one participant declined to participate before treatment started. And no participants were enrolled in Arm C.
Arm/Group | Arm A, Cohort 1 Bintrafusp Alfa (M7824) 1200 mg (Days 1, 15) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1)
All-Cause Mortality (participants affected / at risk) | 2/14 | 1/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/6 | 0/0
Other Adverse Events (participants affected / at risk) | 14/14 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Cohort 1 Bintrafusp Alfa (M7824) 1200 mg (Days 1, 15) (N=14) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) (N=6) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1) (N=0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | NA
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Cohort 1 Bintrafusp Alfa (M7824) 1200 mg (Days 1, 15) (N=14) | Arm B,Cohort 1 M7824 1200mg+TriAdVaccine 5x10e^11viral Particles(ETBX-011,ETBX-051&ETBX-061) (Day 1) (N=6) | Arm C, Cohort 1 M7824 1200mg + TriAd Vaccine 5x10e^11 Viral Particles (Day 1)+N-803 15mcg/kg (Day 1) (N=0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | NA
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | NA
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | NA
Anemia (Blood and lymphatic system disorders) | 3 (4) | 3 (9) | NA
Aphonia (Nervous system disorders) | 1 (1) | 1 (1) | NA
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | NA
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | NA
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | NA
CPK increased (Investigations) | 1 (1) | 0 (0) | NA
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Creatinine increased (Investigations) | 2 (2) | 0 (0) | NA
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | NA
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1) | NA
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | NA
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | NA
Dysphagia (Gastrointestinal disorders) | 4 (5) | 2 (2) | NA
Edema limbs (General disorders) | 1 (1) | 0 (0) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | NA
Eye disorders - Other, Anisocoria, left eyelid droop, pupil asymmetry (Eye disorders) | 0 (0) | 1 (1) | NA
Fatigue (General disorders) | 5 (6) | 3 (5) | NA
Fever (General disorders) | 0 (0) | 1 (1) | NA
Flu like symptoms (General disorders) | 1 (1) | 2 (2) | NA
GGT increased (Investigations) | 1 (1) | 0 (0) | NA
Gait disturbance (General disorders) | 2 (2) | 0 (0) | NA
Gastrointestinal disorders - Other, Sialadenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | NA
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | NA
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | NA
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
Injection site reaction (General disorders) | 0 (0) | 5 (5) | NA
Intraoperative head and neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA
Lipase increased (Investigations) | 2 (2) | 1 (1) | NA
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | NA
Lymphocyte count decreased (Investigations) | 5 (5) | 2 (2) | NA
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA
Neck edema (General disorders) | 0 (0) | 1 (1) | NA
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA — Keratoacanthoma, left clavicle/neck
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA — Lichenoid Dermatitis vs. Keratoacanthoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Right hand bump (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
Oral hemorrhage (Gastrointestinal disorders) | 6 (6) | 3 (3) | NA
Oral pain (Gastrointestinal disorders) | 2 (2) | 4 (5) | NA
Pain (General disorders) | 1 (1) | 1 (1) | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | NA
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | NA
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | NA
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | NA
Surgical and medical procedures - Other, erythema at surgical site right neck (Surgical and medical procedures) | 0 (0) | 1 (1) | NA
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | NA
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | NA
Vaccination site lymphadenopathy (General disorders) | 1 (1) | 0 (0) | NA
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Weight loss (Investigations) | 4 (6) | 0 (0) | NA
White blood cell decreased (Investigations) | 2 (2) | 0 (0) | NA
Wound infection (Infections and infestations) | 3 (3) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT04247282/Prot_SAP_002.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT04247282/ICF_001.pdf